CLINICAL TRIAL: NCT06817408
Title: Cell-free DNA Epigenomics to Track the Dynamics of Organ Damage and Immune Exhaustion During Sepsis
Brief Title: Dynamics of Organ Damage and Immune Exhaustion During Sepsis
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Aadel A. Chaudhuri, Associate Professor of Radiation Oncology, Mayo Clinic
Other Study IDs: 24-009707; 7R35GM142710-04 (NIH)
Record Dates: First submitted 2025-01-14; First posted 2025-02-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Sepsis
Keywords: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma, peripheral blood leukocytes, cfDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observation — One additional blood draw in the Emergency Department as part of their standard of care visit.

SUMMARY:
This is a prospective, non-randomized study investigating if organ damage and immune changes can be measured by liquid biopsy NGS through advanced analytical methods.

DETAILED DESCRIPTION:
To determine the sample size needed to derive a signature matrix to identify novel biomarkers in sepsis, investigators performed a mathematical modeling exercise of the lower limits of sensitivity of this liquid biopsy approach. The detection limit of cell-free nucleic acid analysis is determined in part by the number of independent transcripts or "reporters" that are interrogated. Using an established and independently validated binomial model that was previously applied to the prediction of circulating tumor nucleic acid detection limits, investigators estimated the probability of cell-free nucleic acid detection in sepsis patients based on the number of unique tissue-specific reporters (i.e., hepatic transcripts that may reflect disease severity). This yields a result of n=18 per group to achieve 0.90 power at alpha=0.05. The investigators will thus plan to analyze data from n=18 per cell/tissue type to derive the signature matrix for this project.

ELIGIBILITY:
Inclusion Criteria:

• Patients who've developed a shocked state (Hypotension or Lactate grade >4) or Clinical Concern

Exclusion Criteria:

* <18 years of age
* Pregnant Women
* Nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who've developed a shocked state or clinical concern that are going thru the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Survival | From date of patient enrollment until date of death for any cause or up to 1 year after patient enrollment date, whichever comes first.
  Overall survival

SECONDARY OUTCOMES:
ICU Time | Up to 1 year after patient enrollment date
  Time for patient in ICU
Hospital Stay Duration | Up to 1 year after patient enrollment date
  Days
Renal Replacement Therapy | Up to 1 year after patient enrollment date
  If patient needed renal replacement therapy during duration on study.
Ventilator and Vasopressor Free Days | Up to 1 year after patient enrollment date

CONTACTS AND LOCATIONS:
Overall Officials: Aadel A Chaudhuri, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials